CLINICAL TRIAL: NCT06252857
Title: Real-world Evaluation of (Non-invasive) Diagnostic and Treatment Strategies in Low-Risk Basal Cell Carcinoma: a Prospective Cohort Study
Brief Title: Real-world Evaluation of Diagnostic and Treatment Strategies in Low-Risk Basal Cell Carcinoma
Acronym: REDT-BCC
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0356
Record Dates: First submitted 2024-01-18; First posted 2024-02-12 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Basal Cell Carcinoma
Keywords: imiquimod; surgical excision
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Imiquimod Topical — Topical application of imiquimod (once daily, 5 days a week, during 6 weeks) versus surgical excision.
  Other Names: Surgical Excision

SUMMARY:
Basal cell carcinoma (BCC) is the most prevalent form of cancer among the Caucasian population. There are several subtypes of BCC with different clinical characteristics and treatment strategies. Superficial and nodular BCCs are low-risk BCC subtypes. The diagnosis and subtype of BCC can be confirmed by means of punch biopsy, but non-invasive diagnosis by means of Optical Coherence Tomography (OCT) is proven to be a non-inferior alternative diagnostic instrument. Besides, non-invasive topical treatment is recommended as valuable treatment alternative to surgical excision for low-risk BCC.

Since non-invasive diagnosis and treatment for low-risk BCC is being implemented into daily practice, we want to evaluate the real-world effectiveness of different invasive and non-invasive diagnostic and treatment strategies in the management of low-risk BCC. This real-world evidence will enhance our understanding of these management strategies for low-risk BCC in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Diagnosis of low-risk BCC based on CDE with OCT confirmation or with histopathological verification in case OCT diagnosis is doubtful.
* Tumors meeting the criteria for low-risk BCC
* Patient is able to understand the instruction regarding the study participation and application of IMQ treatment

Exclusion Criteria:

* Tumor location in the H-zone of the face or hairy scalp, anogenital area
* Diagnosis of recurrent BCC or previous skin cancer within 2cm of the treatment area
* Strong suspicion/diagnosis of high-risk BCC subtype or other skin condition on OCT or punch biopsy
* Women who are pregnant or breastfeeding
* Previous allergy or intolerance to IMQ
* No concurrent use any other systemic chemopreventive or immunosuppressive medication during the treatment period, 30 days before start and 3 months after the end of treatment
* Limited understanding of the Dutch language and not being able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the outpatient department of MUMC+ with a clinical suspicion for low-risk BCC, who have a final diagnosis of low-risk BCC confirmed by OCT, or by punch biopsy in case uncertainty about diagnosis remains after OCT. Patients will be treated in accordance with standard care: either SE or IMQ. The choice for treatment is based on shared decision making.
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of imiquimod versus surgical excision | 1 year post-treatment
  Treatment success, expressed as the proportion of tumor free patients

SECONDARY OUTCOMES:
Adverse effects | During imiquimod treatment, reported by the patient
  Incidence and severity of adverse effects
Mean treatment compliance for patients in the imiquimod group | During treatment, reported by the patient in a treatment checklist
  In percentages
Cosmetic outcome | 1 year post-treatment
  Patient-reported satisfaction with cosmetic result of treatment area, expressed as mean score on the DASS questionnaire
Patient treatment satisfaction | 1 year post-treatment
  Patient-reported satisfaction with treatment, expressed as the proportion of patients reporting to be satisfied with their treatment on a 4-point Likert-scale.
Cost-effectiveness analysis | 1 year post-treatment
  Cost-effectiveness will be analysed from a health-care perspective: pre-, during and post-treatment costs will be recorded and analysed and compared in both treatment groups using a cost-effectiveness analysis (CEA)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared upon reasonable request